CLINICAL TRIAL: NCT00703495
Title: Validation of Non- Invasive Regional Transcranial Oxygen Saturation (rSO2) by Comparison With Invasive Brain Tissue Oxygenation (PbtO 2) Measurement in Patients With Severe Traumatic Brain Injury
Brief Title: Invasive and Non-Invasive Assessment of Cerebral Oxygenation in Patients With Severe Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Leal Noval, Santiago R., Hospitales Universitarios "Virgen del Rocio"
Other Study IDs: PI 06/2008
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Brain Injuries
Keywords: traumatic; brain injury; brain regional oxygen saturation (rSO2); brain tissue oxygenation (PbtO2); cerebral perfusion pressure (CPP)
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: transcranial oxygen saturation measurement (INVOS Somanetics 5100C) — rSO2 measurement
  Other Names: INVOS Somanetics 5100C

SUMMARY:
The purpose of this study is to investigate the relationship among regional transcranial oxygen saturation (rSO2), brain tissue oxygen pressure (PbtO2) and cerebral perfusion pressure (CPP) in patients with severe traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Experience with rsO2 assessed by near infrared spectroscopy (NIRS) in patients with severe TBI is lacking. Reports about the usefulness of rSO2 are contradictory as regards its technical reliability and clinical value. Continuous time-domain analysis comparing rSO2, PbtO2 and CPP has never been carried out and the correlation among these variables remains largely unknown. A significant association between rSO2 and these clinically important variables would suggest that cerebral oximetry provides relevant data signifying that rSO2 might be a useful tool assessing cerebral oxygenation in selected patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

* Severe Traumatic Brain Injury (Glasgow Coma Scale < 9)
* Having an intraparenchymal cerebral ICP/PbtO2 catheter previously inserted.
* Expected length of ICU stay > 1 days

Exclusion Criteria:

* Patient's relatives refusal to patient's inclusion in the study
* Patients necessitating ongoing resuscitation
* End-stage in which death is imminent
* Deficient signal of rSO2 impeding its proper valuation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stable patients with severe traumatic brain injury (Glasgow Coma Scale < 9) monitored through intracranial pressure (ICP) and brain tissue partial pressure of oxygen (PbtO2) probe, inserted for indications other than inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
correlation between rSO2 and PbtO2 | four months

SECONDARY OUTCOMES:
correlation between rSO2 and CPP | four months

CONTACTS AND LOCATIONS:
Overall Officials: Santiago R Leal-Noval, M.D., PhD, Principal Investigator — Hospital Universitario "Virgen del Rocío", Seville, Spain; Aurelio Cayuela, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Victoria Arellano, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Yael Corcia, M.D., Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Vicente Padilla, M.D., Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Claudio Garcia-Alfaro, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Antonio Marín, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Francisco Murillo, M.D., PhD, Study Director — Hospital Universitario "Virgen del Rocío", Seville, Spain; Rosario Amaya, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain; Maria Dolores Rincón, M.D., PhD, Study Chair — Hospital Universitario "Virgen del Rocío", Seville, Spain
Locations (1):
- Hospital Universitario "Virgen del Rocío", Seville, Seville, Spain

REFERENCES:
- [Derived] Leal-Noval SR, Cayuela A, Arellano-Orden V, Marin-Caballos A, Padilla V, Ferrandiz-Millon C, Corcia Y, Garcia-Alfaro C, Amaya-Villar R, Murillo-Cabezas F. Invasive and noninvasive assessment of cerebral oxygenation in patients with severe traumatic brain injury. Intensive Care Med. 2010 Aug;36(8):1309-17. doi: 10.1007/s00134-010-1920-7. Epub 2010 May 26. PMID 20502869